CLINICAL TRIAL: NCT04582149
Title: Wearable Eye-Tracking Device as Means of Communication in the Critically Ill and Mechanically Ventilated Patient
Brief Title: Eye-Control Trial: Wearable Eye-Tracking Device as Means of Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Eyefree Assisting Communication Ltd (Industry)
Responsible Party: Principal Investigator, Ofer Sadan, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00114955
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Failure Requiring Mechanical Ventilation
Keywords: Critical illness; Communication; Intensive care unit; Mechanical ventilation
MeSH Terms: conditions — Critical Illness; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- EyeControl Eye-tracking Device (Experimental): Ventilated ICU patients using the EyeControl wearable, eye-tracking device.
  Interventions: Device: EyeControl Eye-tracking Device

INTERVENTIONS:
Device: EyeControl Eye-tracking Device — The EyeControl is a new, wearable, eye-tracking device that facilitates communication by means of internal feedback to the patients with a bone-conducting speaker. In this way, the device can ask the patient what he or she wants to say, and the patient replies by eye gestures such as blinking or moving the eyes in a certain direction. Once the patient is able to operate the device, it will stay on the patient for as long as she or he would like it on, or until the patient is successfully extubated or discharged from the ICU, whichever is earliest.

SUMMARY:
The purpose of this study is to evaluate the feasibility of use of a wearable communication device for critically ill patients who are admitted to the intensive care unit (ICU) and mechanically ventilated. The study will assess the safety, tolerability, and ease of use of the EyeControl device, and examine its potential monitoring capabilities.

DETAILED DESCRIPTION:
Critically ill patients, who are mechanically ventilated, suffer not only from their acute, potentially devastating illness, but also from the lack of ability to communicate in an effective manner. This is the direct result of the orotracheal tube or tracheostomy required for the mechanical ventilation, which does not allow speech to be produced. On top of the mechanical change in air flow, communication challenges result from sedation, neurological injuries (primary brain injury or secondary encephalopathy), and delirium.

Lack of communication can lead to increased frustration, anxiety, and overall psychological stress and could continue to the development of post-traumatic stress disorder (PTSD). On top of the subjective discomfort, the inability to communicate in an effective manner may impair medical care-for example, by failure to assess symptoms such as pain or breathing discomfort by behavioral cues only.

Currently, the solutions for communication deficits in mechanically ventilated patients are mainly using yes/no communication, attempting to write, and communication boards that allow people to point at defined pictures or letters. Recently, technological advancements led to incorporation of more sophisticated communication devices, proving the feasibility of an eye-tracking approach, for example.

The EyeControl is a new, wearable, eye-tracking device that facilitates communication by means of internal feedback to the patients with a bone-conducting speaker. In this way, the device can ask the patient what he or she wants to say, and the patient replies by eye gestures such as blinking or moving the eyes in a certain direction. This approach eliminates the need for calibration, as most eye-tracking devices that use a screen require, and is relatively easy to operate.

This study will assess the safety, tolerability, and ease of use of the EyeControl device.

ELIGIBILITY:
Inclusion Criteria:

* Intensive Care Unit (ICU) Admission
* Mechanically ventilated for at least 24 hours
* Richmond Agitation Sedation Score (RASS) between -1 to 1 at the time of screening
* Ability to follow simple commands

Exclusion Criteria:

* Inability to follow commands during screening (at a minimum: open and close eyes, move eyes to one side or the other)
* Known cerebral injury (acute or chronic) in the dominant hemisphere concerning for aphasia on clinical assessment
* Significant pre-existing neurologic (i.e., dementia and/or cognitive deficiencies), psychiatric, or baseline communication challenges that would confound outcomes assessments
* Inability to blink or move eyes for any reason
* Prisoner or incarceration
* Inability or unwillingness to provide informed consent
* Unwillingness to be contacted for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Sadan, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results reported in the study publications (text, tables, figures, and appendices) will be available for sharing with other researchers, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data will be available for sharing beginning one year after article publication, with no end date.
Access Criteria: Non-study investigators and researchers (i.e., external) may submit their proposal to the study investigators for approval of methodologically appropriate proposals and inquiry. Data will be available for sharing in order to achieve aims in the approved proposal. Proposals should be submitted to the PI at ofer.sadan@emory.edu. Requestors will be required to execute a data use/transfer agreement to receive a limited dataset. Data will be provided directly to external investigators.

REFERENCES:
- [Result] Sadan O, Ratcliff JJ, Samuels OB, Hall AJ. A pilot study to assess the safety and feasibility of a wearable communication device in mechanically ventilated critically ill patients. J Crit Care. 2026 Feb;91:155259. doi: 10.1016/j.jcrc.2025.155259. Epub 2025 Sep 13. PMID 40946530

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University Hospital in Atlanta, Georgia, USA. Participant enrollment began May 19, 2021 and all study assessments were completed by January 23, 2023.
Groups:
- EyeControl Eye-tracking Device: Ventilated ICU patients using the EyeControl wearable, eye-tracking device. The EyeControl is a new, wearable, eye-tracking device that facilitates communication by means of internal feedback to the patients with a bone-conducting speaker. In this way, the device can ask the patient what he or she wants to say, and the patient replies by eye gestures such as blinking or moving the eyes in a certain direction. Once the patient is able to operate the device, it will stay on the patient for as long as she or he would like it on, or until the patient is successfully extubated or discharged from the ICU, whichever is earliest.
Period: Overall Study
Arm/Group | EyeControl Eye-tracking Device
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EyeControl Eye-tracking Device
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 52 [25 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
ICU Type [Count of Participants; unit: Participants]
  Surgical | 12
  Medical | 13
  Neuroscience | 5
Sequential Organ Failure Assessment (SOFA) Score at Admission [Median (Full Range); unit: score on a scale] — The SOFA score is a mortality prediction score that is based on the degree of dysfunction of 6 organ systems (respiratory, nervous, cardiovascular, liver, coagulation, and kidneys). Each organ system is scored on a 5-point scale where normal = 0 and high degree of disfunction = 4. The total score ranges from 0 to 24 and a higher score indicating greater severity. A score of 0-6 is associated with a mortality rate of less than 10% while a score between 16 and 24 is associated with a greater than 90% mortality rate.
  score on a scale | 6 [0 to 15]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) is calculated as weight in kilograms (kg) divided by the square of the body height measured in meters (m). A BMI between 18.5 and 24.9 is considered to be normal weight. A BMI of 25-29.9 indicates overweight, while a BMI of 30 or more indicates obesity.
  kg/m^2 | 28.7 (8.5)
Experienced delirium during admission [Count of Participants; unit: Participants] | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Succeeded in Operating the EyeControl Device
Description: Successful operation of the device was defined as completing a set of assignments termed as a proficiency test. This proficiency test included the ability to call for help and the ability to choose a correct answer out of multiple choice questions that were read to the patient using the device. Participants were able to try to learn to operate the device once per day for up to three days.
Time Frame: Up to Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | EyeControl Eye-tracking Device
Number analyzed (Participants) | 30
Participants | 11

2. Primary Outcome: Time To Successful Operation of the EyeControl Device
Description: Successful operation of the device was defined as completing a set of assignments termed as a proficiency test. This proficiency test included the ability to call for help and the ability to choose a correct answer out of multiple choice questions that were read to the patient using the device. Participants were able to try to learn to operate the device once per day for up to three days. The time (in minutes) of training required for a patient to successfully operate the device was documented.
Time Frame: Up to Day 3
Population: The population in this analysis includes the 11 participants who were able to successfully operate the device.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | EyeControl Eye-tracking Device
Number analyzed (Participants) | 11
minutes | 11 (3)

3. Primary Outcome: Number of Participants Successfully Operating the EyeControl Device Per Attempt Day
Description: Successful operation of the device was defined as completing a set of assignments termed as a proficiency test. This proficiency test included the ability to call for help and the ability to choose a correct answer out of multiple choice questions that were read to the patient using the device. Participants were able to try to learn to operate the device once per day for up to three days. The study day when participants passed the proficiency test was documented.
Time Frame: Up to Day 3
Population: The population in this analysis includes the 11 participants who were able to successfully operate the device.
Measure: Count of Participants; unit: Participants
Arm/Group | EyeControl Eye-tracking Device
Number analyzed (Participants) | 11
Participants
  Day 1 | 8
  Day 2 | 3
  Day 3 | 0

4. Secondary Outcome: Days of Use
Description: The duration of EyeControl device use and participation in the trial was recorded in days (participation in the trial ended when use of the device ended). Participants left the trial due to inability to operate the device, patient request, technical issues, and no longer needing the device (extubation, ICU discharge).
Time Frame: Up to end of study participation (up to 3 days)
Measure: Median (Full Range); unit: days
Arm/Group | EyeControl Eye-tracking Device
Number analyzed (Participants) | 30
days | 1 [1 to 3]

5. Post Hoc Outcome: Clinical Characteristics of Participants Who Passed or Did Not Pass The Proficiency Test
Description: Participants were stratified based on whether or not they passed the proficiency test and were able to successfully operate the EyeControl device. Clinical characteristics (tracheostomy, delirium, and exposure to certain medications) of these groups of participants were examined.
Time Frame: Up to Day 3
Measure: Count of Participants; unit: Participants
Groups:
- Passed Proficiency Test: Study participants who passed the proficiency test and successfully operated the EyeControl device.
- Did Not Pass Proficiency Test: Study participants who did not pass the proficiency test for successfully operating the EyeControl device.
Arm/Group | Passed Proficiency Test | Did Not Pass Proficiency Test
Number analyzed (Participants) | 11 | 19
Participants
  Tracheostomy | 3 | 8
  Delirium detected on day of device use | 1 | 3
  Exposure to fentanyl on day of attempt to use device | 2 | 6
  Exposure to any benzodiazepine on day of attempt to use device | 0 | 1
  Exposure to dexmedetomidine on day of attempt to use device | 6 | 7
  Exposure to propofol on day of attempt to use device | 0 | 2
  Exposure to any pressors on day of attempt to use device | 4 | 3

6. Post Hoc Outcome: SOFA Score of Participants Who Passed or Did Not Pass The Proficiency Test
Description: Participants were stratified based on whether or not they passed the proficiency test and were able to successfully operate the EyeControl device. The Sequential Organ Failure Assessment (SOFA) Score at admission of these groups of participants was compared. The SOFA score is a mortality prediction score that is based on the degree of dysfunction of 6 organ systems (respiratory, nervous, cardiovascular, liver, coagulation, and kidneys). Each organ system is scored on a 5-point scale where normal = 0 and high degree of disfunction = 4. The total score ranges from 0 to 24 and a higher score indicating greater severity. A score of 0-6 is associated with a mortality rate of less than 10% while a score between 16 and 24 is associated with a greater than 90% mortality rate.
Time Frame: Up to Day 3
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Passed Proficiency Test | Did Not Pass Proficiency Test
Number analyzed (Participants) | 11 | 19
score on a scale | 7 [0 to 15] | 4 [0 to 15]

7. Post Hoc Outcome: Age of Participants Who Passed or Did Not Pass The Proficiency Test
Description: Participants were stratified based on whether or not they passed the proficiency test and were able to successfully operate the EyeControl device. The mean age at admission of these groups of participants was compared.
Time Frame: Up to Day 3
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Passed Proficiency Test | Did Not Pass Proficiency Test
Number analyzed (Participants) | 11 | 19
years | 51.9 (15.2) | 50.4 (14.8)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time patients gave consent to participate and continued up to extubation, ICU discharge, or when the participant wanted to stop using the device (up to 3 days).
Description: Adverse events that were potentially related to study activities were collected.
Arm/Group | EyeControl Eye-tracking Device
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EyeControl Eye-tracking Device (N=30)
Transient redness of the skin where device touches the skin (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT04582149/Prot_SAP_000.pdf